CLINICAL TRIAL: NCT03095833
Title: Food Decisions and Reward System: Modulation by Olfaction and Taste
Brief Title: Food Intake Decisions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient on-site staff to manage study
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0681
Record Dates: First submitted 2017-03-24; First posted 2017-03-30 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Healthy
MeSH Terms: interventions — Odorants; Photic Stimulation; Hematologic Tests; Surveys and Questionnaires; Imaging, Three-Dimensional; Genotype

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Influence of cognitive biases on food intake (Other): Determine how high-level cognitive control can affect the price to pay for a food and the olfactory and visual perception of these foods in healthy subjects and Prader-Willi patients.
  Interventions: Other: Odors; Other: Visual stimulation; Other: Experimental Task; Other: Blood tests; Other: Questionnaires and test administered; Other: fMRI
- Modulation of the floral flavor of a wine (Other): Highlight the brain regions involved in the visual bias related to the intensity of a wine's dress combined with the floral character evaluation of its flavor.
  Interventions: Other: Blood tests; Other: Questionnaires and test administered; Other: fMRI; Other: Odors 2; Other: Images; Other: Experimental Task fMRI; Other: Genotyping for susceptibility to β-ionone; Other: Experimental Task 2

INTERVENTIONS:
Other: Odors — Four odors are available: "milk chocolate", "dark chocolate", "pineapple" and "apricot".
  In addition, a neutral odor will be used "clean air", a control odor transmitted during the task by the olfactometer in the same way as the other 4 odors, the only variant being that no odor will be deposited in the U-tube containing the smells. The images corresponding to the odors will be displayed after the odor has been proposed.
  Arms: Influence of cognitive biases on food intake
Other: Visual stimulation — Concerning behavioral passes, the subjects will be in front of a computer screen on which the task will be presented. For fMRI passes, the visual stimulation of the participant is done by a mirror system placed about 10 cm from the participant's eyes, allowing him to watch a translucent screen on which the visual stimuli are projected. The latter have an intensity similar to that of television images, and therefore below the maximum permitted by labor legislation. The stimuli will be projected via a video projector located at the back of the imager.
  Arms: Influence of cognitive biases on food intake
Other: Experimental Task — The olfactory sensitivity and the olfactory identification capacities of the subjects will be evaluated using the ETOC test. Subjects will have to define his state of hunger/satiety thanks to a questionnaire of hunger. Finally, subjects should assess the hedonic nature of the odor and the edibility of the odor source. The task to be performed will be the same for the behavioral study as for the imaging study. The subject will receive instruction from the following three: "indulge yourself", the subject must think of the desire to eat the food that will be presented to him in olfactory and visual form; "Be natural," the subject must act as naturally as possible; Or "hold back," the subject must distance themselves from their desire to eat and control themselves. In a second step, an odor will be presented for 5 seconds. This will be based on the subject's inspiration, then an image associated with the odor will be presented for two seconds.
  Arms: Influence of cognitive biases on food intake
Other: Blood tests — Before and after the imaging examination, a blood sample will be taken by a medical imaging manipulator affiliated with the CERMEP whose actions will be remunerated in accordance with the usual hygiene and safety rules. The samples taken will then be annotated with the subject code and kept at the CERMEP. The volume of ghrelin sampling is 5 ml (10 ml for two samples). The volume of the leptin is 5 ml (ie 10 ml for two samples).
Other: Questionnaires and test administered — The proposed questionnaires respond to all ethical aspects established by international and national standards to undertake studies on human subjects. Two types of questionnaires will be used in this experiment: Inclusion of the Subjects and Exploratory Tests.
Other: fMRI — The purpose of the imaging part is to determine how high-level cognitive control (the setpoint) can affect the price of a food and the olfactory and visual perception of these foods in healthy subjects and Prader-Willi patients.
Other: Odors 2 — To modify the floral character of the wine used, the investigators will use the β-ionone odorant molecule (4 (2,6,6-trimethyl-1-cyclohexenyl) -3-buten-2-one (CAS number 14901-07-6) Purity ≥97.0% (Fluka) This molecule is commonly found in wines with a violet odor.
  Arms: Modulation of the floral flavor of a wine
Other: Images — The visual stimulation of the subject will be done by a system of mirrors placed about 10 cm from the subject's eyes allows him to look at a translucent screen behind the MRI scanner and on which the visual stimuli are projected.
  Arms: Modulation of the floral flavor of a wine
Other: Experimental Task fMRI — For each test the subjects will receive at the same time an image on the screen and a sample of wine (2 ml) delivered in the mouth of the subject thanks to the system of programmable pumps.
  Arms: Modulation of the floral flavor of a wine
Other: Genotyping for susceptibility to β-ionone — Sampling will be done by the subject himself by scratching and firmly pressing into the oral cavity, specifically at the cheeks and tongue for one minute, being careful not to touch the teeth and gums.
  Arms: Modulation of the floral flavor of a wine
Other: Experimental Task 2 — The investigators will determine how perceptual judgments are modulated by cross-modal stimuli, as well as metacognitive judgments (how individuals judge their own sensory performance). In addition, they will determine how perceptual judgments are modified in the context of group decisions and how language influences performance.
  Arms: Modulation of the floral flavor of a wine

SUMMARY:
Functional Magnetic resonance study on the effect of cognitive context variables on the perception and valuation of food odorants and flavor. The study is composed of two experiments; in a first experiment we address the question of how valuation of food odors are modulated by 3 cognitive conditions (indulgence, healthy, and neutral). Food odors are delivered using a custom-made olfactometer. Here we hypothesize that cognitive regulation can modulate the primary sensory processing of food odors. We expect that cortical regions related with valuation and cognitive regulation such as the ventromedial prefrontal cortex and the dorsolateral prefrontal cortex operate the modulation of primary olfactory cortex and amygdala. In a second experiment, we aim to reveal the brain areas involved in integrating food color cues with odor and taste stimuli. Here we hypothesize that color cues are capable of biasing flavor attributes of food (flavor intensity), and that this bias occurs at different cortical areas commonly associate with multisensory integration such as the orbitofrontal cortex, insula, amygdala and hippocampus.

ELIGIBILITY:
Inclusion Criteria:

* healthy or Prader-Willi
* right handed

Exclusion Criteria:

* Nursing or pregnant women
* undergoing medical treatment
* Having known olfactory disorder
* neurological or psychiatric history
* all pertinent conditions according to the use of magnetic resonance imaging.
* anosmia (partial/total)
* neurological, psychological or other disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2015-02-27 (Actual); Primary Completion 2015-11-19 (Actual); Study Completion 2015-11-19 (Actual)

PRIMARY OUTCOMES:
brain activity related to the perception of food odors and flavor | Hour 1
  functional magnetic resonance imaging data

SECONDARY OUTCOMES:
behavioral ratings of odor/flavor valuation by participants | Hour 1
  behavioral ratings of odor/flavor valuation by participants
blood alcohol level post experiment | 10 minutes
  reference value for file information

CONTACTS AND LOCATIONS:
Overall Officials: Caroline DEMILY, MD, Principal Investigator — CH le Vinatier
Locations (1):
- CH le Vinatier, Bron, France